CLINICAL TRIAL: NCT00406445
Title: Metabolic Regulation by Tumor Suppressor p53 in Li-Fraumeni Syndrome
Brief Title: Role of p53 Gene in Metabolism Regulation in Patients With Li-Fraumeni Syndrome
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070030; 07-H-0030
Record Dates: First submitted 2006-11-25; First posted 2006-12-04 (Estimated); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Mitochondrial Disorders; Li-Fraumeni Syndrome; Carriers of p53 Mutation
Keywords: p53 Mutation; Li-Fraumeni Syndrome; Aerobic Metabolism; Magnetic Resonance Spectroscopy
MeSH Terms: conditions — Mitochondrial Diseases; Li-Fraumeni Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- carrier LFS family members: 96 carrier LFS family members
- non-carrier LFS family members or normal: 60 non-carrier LFS family members or normal
- non-carrier mitochondrial disorder family members or normal controls: 20 non-carrier mitochondrial disorder family members or normal controls
- normal controls for MR spectroscopy study: 30 normal controls for MR spectroscopy study
- subjects with mitochondrial disorders: 20 subjects with mitochondrial disorders

SUMMARY:
This study will examine metabolic and biological factors in people with Li-Fraumeni syndrome, a rare hereditary disorder that greatly increases a person's susceptibility to cancer. Patients have a mutation in the p53 tumor suppressor gene, which normally helps control cell growth. This gene may control metabolism as well as cancer susceptibility, and the study findings may help improve our understanding of not only cancer but also other conditions, such as cardiovascular function.

Healthy normal volunteers and patients with the Li-Fraumeni syndrome and their family members may be eligible for this study. Candidates must be at least 18 years of age, in overall good health and cancer-free within 1 year of entering the study. Participants undergo the following procedures:

* Blood tests for routine lab values and for research purposes.
* ECG and echocardiogram (heart ultrasound) to evaluate heart structure and function.
* Resting and exercise metabolic stress testing: The subject first relaxes in a chair wearing the facemask and then exercises on a stationary bicycle or treadmill while wearing the mask. This test uses the facemask to measure oxygen usage by the body to determine metabolic fitness. Electrodes are placed on the body to monitor the heart in an identical manner to a standard exercise stress test.
* Magnetic resonance imaging of metabolism: The subject lies on a bed that slides into a large magnet (the MRI scanner) for up to 60 minutes. During scanning, the arm or leg muscles are stressed by inflating a blood pressure cuff and by exercising the limb for several minutes. Subjects may be asked to squeeze a rubber ball or exercise with a foot pedal. Immediately afterwards, the pressure in the cuff is released and remains deflated for 10 to 15 minutes. No more than three 5-minute episodes of blood flow stoppage are performed.
* Standard MRI scan of exercised limb to determine muscle volume.
* Brachial artery reactivity test to measure blood vessel function: Before the exercise stress testing, subjects lie on a stretcher while the brachial artery (artery in the forearm) is imaged using a noninvasive ultrasound method. Artery size and blood flow velocity are measured before and after inflating a blood pressure cuff on the forearm. Vessel size and flow velocity measurements are repeated after 15 minutes and again after administration of nitroglycerin under the tongue.
* Oral glucose tolerance testing to test for diabetes: To assess sugar metabolism, subjects drink a sugar solution. Blood samples are collected before drinking the solution and 1 and 2 hours after drinking the solution.
* Muscle biopsy (optional according to subject preference): Subjects may be given small amounts of sedation for the procedure. A small area of skin over a leg muscle is numbed and a small amount of muscle tissue is surgically removed.

DETAILED DESCRIPTION:
We have previously reported that TP53 (encoding p53 protein), one of the most frequently mutated genes in human cancers, dose dependently modulates the balance between the utilization of oxidative and glycolytic pathways for energy generation in human colon cancer cells and mouse liver mitochondria. Though morphologically similar to their wild-type littermates, mice deficient in p53 display a gene dose-dependent decrease in aerobic exercise capacity, implying that p53 has functions beyond its well characterized cell cycle activities. These current findings have broad implications in fields ranging from cancer and aging research to cardiovascular physiology.

In the Li-Fraumeni familial cancer syndrome (LFS), affected individuals harbor a germline mutation in TP53, hence they are heterozygous with reduced wild-type p53 activity. We hypothesize that the heterozygous individuals will display alterations in aerobic capacity and metabolism that previously has been unappreciated. This IRB proposal translates our experimental observation to human subjects in collaboration with extramural groups studying this rare familial syndrome. The results may not only help clarify why mutations of p53 gene are so common in cancers by potentially conferring metabolic advantages in tumorigenesis, but they may also give us an opportunity to understand a fundamental regulatory mechanism in cellular energy generation relevant to other processes.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. At least 18 years of age and able to give informed consent
  2. In overall good physical and mental health;
  3. Able to exercise on a treadmill (if participating in the treadmill exercise portion).
  4. Able to perform hand or leg exercises (if participating in the MRS portion)

Able to undserstand and sign consent

Have been diagnosed with the Li-Fraumeni Syndrome or have a family member with the Li-Fraumeni Syndrome or have been diagnosed with mitochondrial disorder or be a healthy volunteer

EXCLUSION CRITERIA:

Cancer patients undergoing or requiring systemic treatment

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 96 carrier LFS family members 60 non-carrier LFS family members or normal 30 normal controls for MR spectroscopy study 20 subjects with mitochondrial disorders 20 non-carrier mitochondrial disorder family members or normal controls
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2007-01-23 (Actual); Primary Completion 2021-03-22 (Actual); Study Completion 2021-03-22 (Actual)

PRIMARY OUTCOMES:
Non-invasively measure aerobic exercise capacity and metabolism | ongoing
  Because an interim analysis has confirmed our hypothesis, the aim of the primary endpoint has been achieved.

SECONDARY OUTCOMES:
Non-invasively measure markers of mitochondrial function by magneticresonance spectroscopy (MRS) in response to transient ischemic stress | ongoing
  This will serve to facilitate bench-to-bedside studies to investigate metabolic and other associated changes in LFS with the goal of deriving mechanistic insights that may lead to new strategies forcancer prevention.
Measure oxygen consumption, protein and RNA levels of p53-regulated mitochondrial genes using blood cells and other tissue samples if available. | ongoing
  This will serve to facilitate bench-to-bedside studies to investigate metabolic and other associated changes in LFS with the goal of deriving mechanistic insights that may lead to new strategies forcancer prevention.

CONTACTS AND LOCATIONS:
Overall Officials: Paul M Hwang, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Arena R, Myers J, Abella J, Peberdy MA. Influence of heart failure etiology on the prognostic value of peak oxygen consumption and minute ventilation/carbon dioxide production slope. Chest. 2005 Oct;128(4):2812-7. doi: 10.1378/chest.128.4.2812. PMID 16236959
- [Background] Brown BW, Costello TJ, Hwang SJ, Strong LC. Generation or birth cohort effect on cancer risk in Li-Fraumeni syndrome. Hum Genet. 2005 Dec;118(3-4):489-98. doi: 10.1007/s00439-005-0016-x. Epub 2005 Nov 12. PMID 16284780
- [Background] Bergman RN, Phillips LS, Cobelli C. Physiologic evaluation of factors controlling glucose tolerance in man: measurement of insulin sensitivity and beta-cell glucose sensitivity from the response to intravenous glucose. J Clin Invest. 1981 Dec;68(6):1456-67. doi: 10.1172/jci110398. PMID 7033284
- [Derived] Wang PY, Li J, Walcott FL, Kang JG, Starost MF, Talagala SL, Zhuang J, Park JH, Huffstutler RD, Bryla CM, Mai PL, Pollak M, Annunziata CM, Savage SA, Fojo AT, Hwang PM. Inhibiting mitochondrial respiration prevents cancer in a mouse model of Li-Fraumeni syndrome. J Clin Invest. 2017 Jan 3;127(1):132-136. doi: 10.1172/JCI88668. Epub 2016 Nov 21. PMID 27869650
- [Derived] Wang PY, Ma W, Park JY, Celi FS, Arena R, Choi JW, Ali QA, Tripodi DJ, Zhuang J, Lago CU, Strong LC, Talagala SL, Balaban RS, Kang JG, Hwang PM. Increased oxidative metabolism in the Li-Fraumeni syndrome. N Engl J Med. 2013 Mar 14;368(11):1027-32. doi: 10.1056/NEJMoa1214091. PMID 23484829
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2007-H-0030.html